CLINICAL TRIAL: NCT00999011
Title: Dose of Early Therapeutic Mobility: Does Type or Frequency Matter?
Acronym: ETM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Chris Winkelman, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NR10781-01A1; 1R21NR010781-01A1 (NIH)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness
Keywords: critical care; inflammatory biomarkers; cytokines; mechanical ventilation; activity; mobility therapy; More than 48 hours of mechanical ventilation
MeSH Terms: conditions — Critical Illness; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One 20 minute period of activity daily (Active Comparator): passive and/or active range of motion, chair sitting, sitting at edge of bed, standing and walking
  Interventions: Procedure: once daily mobility activity
- Two periods of 20 minute activity daily (Active Comparator): passive and/or active range of motion, chair sitting, sitting at edge of bed, standing and walking
  Interventions: Procedure: twice daily mobility activity

INTERVENTIONS:
Procedure: once daily mobility activity — in bed and out-of-bed activity including range of motion, chair sitting, sitting at edge of bed without weightbearing, standing, walking.
  Arms: One 20 minute period of activity daily
Procedure: twice daily mobility activity — as with once daily. Goal is to progress intensity and duration of activity over time as patient condition improves for both arms
  Arms: Two periods of 20 minute activity daily

SUMMARY:
This study will examine the effects of once and twice daily activity performed with patients who are breathing with the aid of a machine in an intensive care unit. Activity can occur in bed. Activity can include transfer to a chair and even walking once the patient's condition allows safe, out-of-bed activity. The investigators hypothesize that early, progressive activity will reduce inflammatory molecules in the blood, promote muscle and physical health and help patients to recover more quickly from critical illness.

DETAILED DESCRIPTION:
Early therapeutic mobility (ETM) activity has been recommended to facilitate recovery and improve outcomes for the survivors of critical illness who experience prolonged mechanical ventilation. The effective dose (i.e., type, frequency and duration) of ETM activity is not known and there are limited reports about the application and effects of ETM in mechanically ventilated intensive care unit (ICU) patients. Three inflammatory biomarkers, interleukin (IL)-6, IL-10 and C-reactive protein, are potentially altered by a single episode of ETM activity. Systemic markers of physical health (i.e., vital signs, delirium, muscle strength, ventilator associated pneumonia, and duration of mechanical ventilation) may also be positively influenced by ETM. The primary aim of this interdisciplinary study is to compare the immediate effects of frequency--single and twice daily episodes--of ETM activity and the effects of type--low and moderate intensity--of ETM activity on molecular biomarkers of inflammation and systemic markers of physical health in mechanically ventilated adults. This is an experimental design, using repeated measures; subjects will be randomized to receive either one or two episodes of ETM activity daily during week days while in the ICU. Type of activity will be determined by patient condition. The research questions are:

1. a. What are the differences between the frequency (once versus twice daily) of ETM activities on inflammatory biomarkers: interleukin (IL)-6, IL-10 and C-reactive protein (CRP)? 1.b. What are the differences between the type (low or moderate) of ETM activities on inflammatory biomarkers: IL-6, IL-10 and CRP?
2. a. What are the differences between frequency of ETM activities on systemic markers of physical health: vital signs, delirium, muscle strength, ventilator-associated pneumonia and duration of mechanical ventilation? 2.b. What are the differences between type of ETM activities on systemic markers of physical health: vital signs, delirium, muscle strength, ventilator-associated pneumonia and duration of mechanical ventilation?

Data will be collected for a maximum of 3 contiguous days in ICU patients who are mechanically ventilated for >48 hours, then weekly to examine short-term patient responses to ETM activities in this preliminary study. Daily episodes of activity will be provided by a study interventionist. Repeated measures MANCOVA and ANCOVA will be used to answer the research questions. This collaborative study evaluates a biobehavioral methodology within an interdisciplinary team consistent with the biobehavioral methods to improve outcome research (PA-07-008) and the mission of the National Institute of Nursing Research to improve treatments and health based on evidence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who require invasive mechanical ventilation for more than 24 continuous hours in the surgical (SICU) or medical ICU (MICU)
* a P:F ratio > 100
* FiO2 < 60% and PEEP less than 10 cmH20 at baseline
* resting vital signs of HR 50-110, mean arterial pressure (MAP) 60-110 mmHg, peripheral oxygenation saturation (SpO2) greater than 88%. Exclusion Criteria:
* There are no exclusions based on gender or minority status.
* Patients will be excluded if they have pre-existing or current neurological, muscular or orthopedic disorders that require inactivity or immobilization during acute care or experience paresis/paralysis that will not improve. Examples of exclusionary conditions include end-stage muscular dystrophy, myasthenia gravis, new quadriplegia, coma, increased intracranial pressure, unrepaired hip fracture and multiple lower extremity fractures.
* Patients for high risk of death will also be excluded, using criteria established by Norton et al.: ICU admission following a hospital stay of >9 days in the past 12 months; age >80 in the presence of 2 or more life-threatening illnesses (e.g., end-stage renal disease, severe heart failure (HF); diagnosis of an active stage IV malignancy; status post cardiac arrest; and diagnosis of intracerebral hemorrhage requiring mechanical ventilation.[99].
* Subjects over 400 pounds can be excluded from mobilization based on the judgment of the bedside nurse or project manager; if the risk for staff or patient harm from moving a patient with excessive weight is considered likely, mobilization will not occur.
* Criteria for exclusion include inability to stand or walk for at least 10 minutes prior to admission; inability to shift weight in bed or assist with turning, inability of staff to access bariatric equipment such as an overhead trapeze, chair, or walker.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in molecular biomarkers of inflammation day 1 of intervention | 1 day
  IL-6, IL-10, C-reactive protein.
Change in molecular biomarkers of inflammation day 2 of intervention if patient still in ICU | 1 day
  IL-6, IL-10, C-reactive protein.
Change in molecular biomarkers of inflammation day 3 of intervention if patient still in ICU | 1 day
  IL-6, IL-10, C-reactive protein.
Vital Signs included RR, HR, and SBP. Change in Respiratory Rate day 1 of intervention. | Baseline = time during rest immediately preceding the intervention. Intervention = 30 min of activity
  Change is Respiratory rate (RR),measured in breaths per minute, during the intervention and comparing to baseline (rest) only.
Change in Respiratory Rate day 2 of intervention if patient still in ICU. Heart Rate and Systolic Blood Pressure. Each vital sign is measured separately and not aggregated. | Baseline RR = time during rest immediately preceding the intervention. Intervention RR = 30 min activity
  Breaths per minute as recorded on the bedside monitor Change defined as the difference between RR at rest and highest RR during the intervention.
Change in Respiratory Rate day3 of intervention if patient still in ICU. | Baseline RR = time during rest immediately preceding the intervention. Intervention RR= during 30 min of activity
  Breaths per minute as recorded on the bedside monitor Change defined as the difference between RR at rest and RR duriing activity.
Vital Signs. Change in Heart Rate day 1 of intervention | ring rest immediately preceding the intervention. Outcome = highest and lowest values during the mobility intervention.
  Change in Heart rate (HR), measured in beats per minute, during the intervention only comparing to baseline. The bedside ICU monitor was used.
Change in Heart Rate day 2 of intervention if patient still in ICU | Once daily or twice daily for up to 3 days of intervention. Baseline = time during rest immediately preceding the intervention. Outcome = highest and lowest values during the mobility intervention.
  Change in Heart rate (HR), measured in beats per minute, during the intervention only comparing to baseline. The bedside ICU monitor was used.
Change in Heart Rate day 3 if patient still in ICU | Once daily or twice daily for up to 3 days of intervention. Baseline = time during rest immediately preceding the intervention. Outcome = highest and lowest values during the mobility intervention.
  Change in Heart rate (HR), measured in beats per minute, during the intervention only comparing to baseline. The bedside ICU monitor was used.
Vital Signs , Change in Systolic Blood Pressure day 1 | Once daily or twice daily for up to 3 days of intervention. Baseline = time during rest immediately preceding the intervention. Outcome = highest and lowest values during the mobility intervention.
  Change in SBP, measured inmmHg, during the intervention only comparing to baseline. The bedside ICU monitor was used. The highest and lowest values were recorded for analysis. The largest change from baseline rest were used in analysis (Rest - Highest value obtained during intervention. This was done 3 times (once daily for up to 3 days) if randomized to once daily interventions or up to 6 times if randomized to twice daily intervention over 3 days.
Vital Signs. Change in Systolic Blood Pressure day 2 of intervention if patient still in ICU | Once daily or twice daily for up to 3 days on intervention. Baseline = time during rest immediately preceding the intervention Outcome = highest and lowest values during the mobility intervention.
  Change in Systolic blood pressure (SBP), measured in millimeters of mercury (mmHg) during the intervention comparing to baseline. The bedisde ICU monitor was used if an arterial indwelling line was present. An automatic BP cuff (dynometer) was used at the start and every 5 minutes if an indwelling line was used. The highest and lowest values were recorded during the intervention.
Change in Systolic Blood Pressure Day 3 of intervention if patient still in ICU | Once daily or twice daily for up to 3 days on intervention. Baseline = time during rest immediately preceding the intervention Outcome = highest and lowest values during the mobility intervention.
  Change in Systolic blood pressure (SBP), measured in millimeters of mercury (mmHg) during the intervention comparing to baseline. The bedisde ICU monitor was used if an arterial indwelling line was present. An automatic BP cuff (dynometer) was used at the start and every 5 minutes if an indwelling line was used. The highest and lowest values were recorded during the intervention.
The total number of days of Mechanical Ventilation while in the ICU | Measured one time, at the discharge from the ICU
  . This is a one-time value. This is the total number of days the patient received invasive mechanical ventilation as documented in the record.
Muscle strength day 1 | Measured once after the intervention on day 1. Collected as many as 3 times if the patient received 3 days of intervention
  This was measured with hand grip using a dynometer and reported as dynes or kg of force.
Muscle strength day 2 | Measured once after the intervention. Collected as many as 3 times if the patient received 3 days of intervention
  This was measured with hand grip using a dynometer and reported as dynes or kg of force.
Muscle strength day 3 | Measured once after the intervention. Collected as many as 3 times if the patient received 3 days of intervention
  This was measured with hand grip using a dynometer and reported as dynes or kg of force.
Change in muscle strength | Collected once after the interention on days 1, 2, 3. The maximum potential change was defined as Day 1-Day 3 but Day 1 -Day was used for patients who were discharged from the ICU on Day 2 and had no data for Day 3
  This was defined as the difference in dynes from Day 1 to Day 3, if the patient was in the ICU for 3 days, or the change from Day 1 to 2 if in the ICU for only 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris Winkelman, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Frances Payne Bolton School of Nursing Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winkelman C, Sattar A, Momotaz H, Johnson KD, Morris P, Rowbottom JR, Thornton JD, Feeney S, Levine A. Dose of Early Therapeutic Mobility: Does Frequency or Intensity Matter? Biol Res Nurs. 2018 Oct;20(5):522-530. doi: 10.1177/1099800418780492. Epub 2018 Jun 14. PMID 29902939